CLINICAL TRIAL: NCT05560178
Title: The Effect of Sexual Health Education Given to Women in the Postmenopausal Period on Sexual Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Serap Kırıcı, researcher, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUserapkirici
Record Dates: First submitted 2022-09-07; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Sexuality; Menopause; Sexual Behavior
Keywords: sexuality; sexual health; postmenapause
MeSH Terms: conditions — Sexuality; Sexual Behavior | interventions — Sex Education

STUDY DESIGN:
Intervention Model Description: Research, parallel group (experiment-control) randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Since it is not possible to blind the experimental and control groups in the study, only statistical blinding will be applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Training group (Experimental): women in the intervention group will be given sexual health education once a week for 4 weeks
  Interventions: Other: SEXUAL HEALTH EDUCATION
- No Intervention: control group (No Intervention): Women will be monitored without any intervention

INTERVENTIONS:
Other: SEXUAL HEALTH EDUCATION — Women in the intervention group will be given sexual health education once a week for 4 weeks
  Arms: Experimental: Training group

SUMMARY:
With this study, it is aimed to evaluate the effect of sexual health education given to women in the postmenopausal period on sexual myths, sexual distress and sexual quality of life.

Type of Research The study was planned as a parallel group (experiment-control) randomized controlled trial.

DETAILED DESCRIPTION:
Establishment of the Study Group: The Female Sexual Function Index (FSFI) was applied to the women who applied to the Obstetrics and Gynecology outpatient clinics of Karaman Training and Research Hospital to determine the study group, and the women who accepted to participate in the study in accordance with the sample selection criteria were applied to the study. General information about the study will be given and general consent will be taken for participation in the research. Then, the Individual Information Form, Sexual Myths Scale (SMS), Female Sexual Distress Scale (Revised- FSDS-R) and Sexual Life Quality Scale-Female (SILK-F) was applied. In accordance with the sample size determined by power analysis, the experimental and control groups were randomly assigned.

blinding Since it is not possible to blind the experimental and control groups in the study, only statistical blinding applied.

Application Steps of the Research Researcher; By introducing themselves to the experimental and control groups, verbal and written information was given about the subject of the research and the steps to be followed. Then, among the women determined by the researcher in accordance with the sample selection criteria, applications were made to the women who were allocated to the experimental group by randomization, and no intervention was made to those who were allocated to the control group.

For the Experimental Group; Sexual Health Education Program The women in the experimental group were given training in line with the "Sexual Health Education Manual for Postmenopausal Women" prepared by the researchers. The training plan of the research is as follows.

Education Plan (Sexual Health Education) Session Subject

1. Female reproductive organs (Female internal and external reproductive organs and sexual anatomy), Male reproductive organs and sexual anatomy Definitions related to sexuality and sexual health (sexuality, sexual health, sexual intimacy, sexual intercourse, sexual behaviors, sexual function, sexual dysfunction)
2. Sexual myths and taboos, sexual distress, sexual quality of life Female sexual function physiology and sexual response cycle, female sexual dysfunctions
3. Definition of menopause, classification of menopause, factors affecting menopause, the effect of menopause on sexual life, changes in the postmenopausal period and its effect on sexual life
4. Recommendations about changes in the postmenopausal period and sexual problems Kegel exercises, masturbation exercises

For the Control Group; Control Group: No intervention was made after the pre-tests were applied to the control group women. However, after the post-tests were applied, a sexual health education and training booklet was given to the control group, taking into account the right to be informed in terms of ethics.

ELIGIBILITY:
Inclusion Criteria:

* Literate,
* Able to communicate verbally,
* Turkish speaking,
* No hearing or vision loss,
* Voluntarily participated in the research,
* Postmenopausal period,
* Natural menopause,
* no sexual dysfunction,
* be less than 65 years old,
* good sexual function

Exclusion Criteria:

* Hormone replacement therapy
* Early menopause (before age 40)
* A chronic systemic disease and/or a psychiatric health problem
* Any sexual education before or during work
* Sexual dysfunction

Ages: 41 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 124 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-27 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Sexual Myths Scale-SMS | Time Frame: 13 weeks
  It is a scale developed to describe sexual myths. The minimum score obtained from the scale is 28, and the maximum score is 140. The cronbach's alpha coefficient of the scale was found to be 0.91. In addition, the sub-dimensions' item scores can be summed to obtain sub-dimensions' scores. It is not the cut-off point of the scale, and the high score indicates that the sexual myths are high.
  The Sexual Myths Scale-SMS will be used to assess sexual myths in each participant.

SECONDARY OUTCOMES:
Female Sexual Distress Scale-Revised- FSDS- R | Time Frame: 13 weeks
  Female Sexual Distress Scale, Derogatis et al. (2008) to measure personal distress related to sexuality in women with sexual dysfunction.
  Responses to the items on the Likert-type scale consist of never (0), rarely (1), sometimes (2), often (3), or always (4). The lowest score that can be obtained from the FSDS-R is "0" and the highest score is "52". Higher scores indicate higher levels of sexual distress.
  FSDS-R will be used to assess sexual myths in each participant.

OTHER OUTCOMES:
Sexual Quality of Life Questionnaire-Female (SQLQ-F) | Time Frame: 13 weeks
  Symonds et al. It was developed by in 2005 to assess the quality of sexual life in women. The scale is easy to apply, six-point Likert type, which individuals can answer on their own, and consists of 18 items. Each item is expected to be answered considering the sexual life in the last four weeks. A high score from the scale indicates that the quality of sexual life is in good condition. SQLQ-F will be used to assess the quality of sexual life in each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Emel Ege, Professor, Study Director — Necmettin Erbakan University; Serap Kırıcı, Investigator:, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Karamanoğlu Mehmetbey University, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No